CLINICAL TRIAL: NCT01162850
Title: A Randomized Double-Blind Placebo Controlled Study Evaluating the Effectiveness and Tolerability of Oral Polypodium Leucotomos in Patients With Melasma
Brief Title: Oral Polypodium Leucotomos for Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Heather Woolery-Lloyd, MD, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20070050
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2008-07

CONDITIONS: Melasma
Keywords: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polypodium Leucotomos (Active Comparator): Oral Polypodium Leucotomos twice daily plus sunscreen SPF 45 for 12 weeks.
  Interventions: Dietary Supplement: Polypodium Leucotomos
- Placebo (Placebo Comparator): Oral Placebo twice daily plus sunscreen SPF 45 for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Polypodium Leucotomos — Oral capsule at 240 mg taken twice a day for 12 weeks
  Arms: Polypodium Leucotomos
Dietary Supplement: Placebo — 240 mg Placebo taken orally twice daily created by company which manufactured active ingredient
  Arms: Placebo

SUMMARY:
Primary Objective: To determine whether there is improvement in the melasma of participants taking oral Polypodium Leucotomos Secondary Objective: To determine whether oral Polypodium Leucotomos is well tolerated in study subjects with melasma.

To determine whether treatment with Polypodium Leucotomos improves the health-related quality of life.

DETAILED DESCRIPTION:
Polypodium Leucotomos is a fern, also known as Calaguala used by the natives of northern Honduras as a treatment against malignant tumors Used in Spain and Central America for the treatment of psoriasis, atopic dermatitis and repigmentation of vitiligo.

Oral Polypodium Leucotomos is safe and effective in patients with melasma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects 18-50 years of age.
* Female subjects with epidermal melasma.
* Female subjects of child-bearing potential must have been willing to use an acceptable form of birth control for the duration of the study.
* Subjects with Fitzpatrick skin types II, III, & IV
* Subjects enrolled in this trial had a 2 week washout period if on prior treatment for melasma.

Exclusion Criteria:

* Pregnant or lactating
* Dermal Melasma
* Hormonal therapies less than or equal too 4 weeks prior to study
* Use of photosensitizing medications
* Simultaneous use of any form of treatment for melasma
* Subjects who were concurrently receiving light therapies
* Subjects who were unwilling to limit the amount of sun exposure
* Simultaneous ( or past 30 day) participation in a clinical research study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Melasma Area and Severity Index (MASI) | Day 0, Week 4, Week 8, Week 12
  The following equation is used to determine the MASI score: MASI = .3A(D+H) [forhead] + .3A(D+H)[right malar] + .3A(D+H)[left malar] + .1A(D+H)[chin]; A = area, D = darkness, and H = homogeneity. Area is based on percentage of the region covered by melasma using a 1-6 scale. Darkness is determined on a 0-3 scale. Homogeneity is based on a 0-4 scale.

SECONDARY OUTCOMES:
Patient Assessment | Week 4, Week 8, Week 12
  Subject critiqued their melasma as either getting worse, showing no improvement, mild improvement or as showing marked improvement upon using the treatment.
Evaluation of Photographs | Post-Week 12
  Photos were evaluated using the grading of worse, no improvement, mild improvement or marked improvement comparing week 12 to baseline.
Adverse Events | Week 4, Week 8, Week 12
  Recorded any and all adverse events that occurred even if it was unlikely that it was associated with the study product.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Woolery-Lloyd, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Cosmetic Center, Miami, Florida, United States